CLINICAL TRIAL: NCT06608771
Title: Implementation of the New Guidelines on the Management of Patients Resuscitated From Cardiac Arrest and Impact on Survival: a Multicenter Retrospective Observational Study
Brief Title: Outcome of Cardiac Arrest Patients Following Guidelines Implementation Over the Years
Acronym: IMPACT-ACC
Status: Recruiting | Type: Observational
Sponsor: Mauro Panigada (Other)
Responsible Party: Sponsor-Investigator, Mauro Panigada, Medical Doctor, Head of the Intensive Care Unit, Department of Anaesthesia, Intensive Care and Emergency, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Policlinico Hospital
Organization: Policlinico Hospital (Other)
Other Study IDs: 5033
Record Dates: First submitted 2024-08-08; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; In-Hospital Cardiac Arrest; Guidelines Implementation; Resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest (OHCA) and In-hospital cardiac arrest (IHCA) patients: The study population includes all adult patients resuscitated from cardiac arrest and subsequently admitted to the Intensive Care Unit over a 14-year-period

SUMMARY:
The study aims to evaluate the level of local implementation of the new interventions introduced by the guidelines for post-cardiac arrest management and their impact on the survival of patients resuscitated from cardiac arrest and admitted to intensive care over a 14-year period. During this time period, the European Resuscitation Council (ERC) and the European Society of Intensive Care Medicine (ESICM) introduced three new guidelines for post-cardiac arrest management, each five years apart: the 2010, 2015, and 2021 guidelines.

DETAILED DESCRIPTION:
This study is a retrospective multicenter cohort observational study (two centers involved: Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico and Fondazione IRCCS San Gerardo dei Tintori).

All patients admitted to the Intensive Care Units (ICU) of the hospitals involved in the study from January 1, 2011, to May 30, 2024, following cardiac arrest of any etiology, who meet the inclusion and exclusion criteria, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients resuscitated from cardiac arrest and admitted to intensive care unit
* Age ≥ 18 years
* Out-of-hospital and in-hospital cardiac arrest
* Cardiac arrest of any etiology

Exclusion Criteria:

* Pediatric patients (<18 years)
* Patients not admitted to one of the aforementioned intensive care units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients resuscitated from cardiac arrest and admitted to ICU over a 14-year-period
Sampling Method: Probability Sample
Enrollment: 693 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit (ICU) Survival | From cardiac arrest date to ICU discharge or death, up to 90 days
  To evaluate ICU survival for patients resuscitated from cardiac arrest
Neurological recovery at ICU discharge | From cardiac arrest date to ICU discharge or death, up to 90 days
  ICU Survival with Cerebral Performance Category (CPC) score of 1 or 2

SECONDARY OUTCOMES:
Hospital discharge status | From cardiac arrest date to hospital discharge or death, up to 180 days
  To evaluate hospital survival for patients resuscitated from cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Ristagno, MD, PhD, Principal Investigator — IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (2):
- Italy (2):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan

IPD SHARING:
Plan to Share IPD: No